CLINICAL TRIAL: NCT03528148
Title: China Medical University Hospital Asia University Hospital
Brief Title: The Effects of Elliptical Cross Training Bike for Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Attending physician,rehabilitation department, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH107-REC2-026
Record Dates: First submitted 2018-04-21; First posted 2018-05-17 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Stroke
Keywords: Post stroke; Gait; Elliptical cross bike.; Postural control; Balance
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomize control trials
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active cycling group (Experimental): effect of combine cycling and conventional physical therapy in quality of life, functional activity and ADL, postural control, balance, muscle tone, spasticity, motor functioning, gait of stroke patients.
  Interventions: Behavioral: cycling; Behavioral: Physical therapy
- control group (Active Comparator): effect of combine conventional physical therapy in quality of life, functional activity and ADL, postural control, balance, muscle tone, spasticity, motor functioning, gait of stroke patients.
  Interventions: Behavioral: Physical therapy

INTERVENTIONS:
Behavioral: cycling — Active cycling
  Arms: active cycling group
Behavioral: Physical therapy — Conventional physical therapy

SUMMARY:
To investigate the effects of elliptical cross bike exercises combine conventional physical therapy on gait, postural control, balance, muscle tone, spasticity, quality of life, motor functioning, functional activity, and ADL in post stroke patients.

DETAILED DESCRIPTION:
In a single-blind, randomized controlled intervention, patients were randomly assigned to an active cycling group (ACG, n=25) five times a week combine with conventional al physical therapy or a control group (CG, n=25) with conventional physical therapy 3 weeks of training in the center.

All outcome measures were administered at the beginning of the study, at the end of the 1st, 2nd, and 3rd week.

All participants will be divided two groups. One group will be experiment with conventional physical therapy as control group (CG), the other group will active cycling as active cycling group (ACG) with elliptical Cross Trainer & Exercise Bike after conventional physical therapy.

Baseline assessment of muscle tone by Myoton-3, Modified Ashworth Scale used as a simple measure of spasticity; Barthel Index scale for performance in activities of daily living; Berg Balance Scale to measure balance; the upper and lower limb subscale of the Fugl-Meyer assessment for motor function of extremities; and BTS G-WALK was used to measure gait parameters. The data will be collect before session.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke (World Health Organization ,1978).
* Joint mobility ranges of lower extremity that would not preclude pedaling(Ambrosini, Ferrante et al. 2011).
* Unilateral hemiplegia.
* Able to carry out simple instructions.
* Able to sit independent at least 20 minutes and pedal an elliptical cross bike.

Exclusion Criteria:

* Neurologic disorders with impaired functionality existing pre-stroke.
* Patients could not follow instructions.
* Cardiovascular disease or other risk factor which precluded participation in aerobic exercise.
* Peripheral neuropathy that could potentially interfere with this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-03-13 (Estimated); Study Completion 2019-03-13 (Estimated)

PRIMARY OUTCOMES:
Gait | 3 weeks
  Subjects were asked to walk at a self-selected speed using walking aids if necessary with 10 m. BTS G-WALK was used to measure characterized of the hemiparetic gait such as speed, cadence and step length of the stroke patients

CONTACTS AND LOCATIONS:
Overall Officials: Chou Li-Wei, PhD, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No